CLINICAL TRIAL: NCT02095912
Title: Aggressive Squamous Cell Carcinoma in Organ Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-2013-0591
Record Dates: First submitted 2014-02-18; First posted 2014-03-26 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Squamous Cell Carcinoma
Keywords: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To identify risk factors for aggressiveness in Squamous Cell Carcinoma of the skin in organ transplant recipients.

DETAILED DESCRIPTION:
Squamous Cell Carcinomas (SCC) are one of the most common skin cancers. They belong to the epithelial neoplasm of the skin, which manifest a local aggressive growth and have potential for metastasis. Organ transplant recipients have a hundredfold higher incidence of SCC.

Unfortunately the primary tumor, regional nodes, metastasis (TNM)-Classification for the prognosis of SCC in this group of patient has not yet been established. Therefore there are no standardised criteria for evaluation of local recurrence or prognosis.

The aim of this study is to identify criteria, which permit a risk assessment relating to aggressiveness of SCC.

ELIGIBILITY:
Inclusion Criteria:

Organ transplant recipients with:

* > 9 SCC in total or
* > 2 SCC per year (in any one year) or
* any single "index" SCC that has a very poorly differentiated cell morphology or that behaved aggressively in Terms of local recurrence or local/systemic metastasis

Exclusion Criteria:

* Non organ transplant recipients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Organ Transplant Recipients with:
  * > 9 Squamous Cell Carcinoma (SCC) in total or
  * > 2 SCC per year (in any one year) or
  * any single "index" SCC that has a very poorly differentiated cell morphology or that behaved aggressively in Terms of local recurrence or local/systemic metastasis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Diameter of Squamous Cell Carcinoma | 1 year
  * Location
  * exact size in mm
  * histological classification (well-differentiated, moderately-differentiated, poorly differentiated, spindle cell morphology, desmoplastic, basi-squamous, acantholytic)
  * Invasion
  * rapid growth
  * local recurrence
  * sentinel node sampling
  * Metastasis

SECONDARY OUTCOMES:
Sun exposure history | 1 year
  * skin type
  * hair colour
  * eye colour
  * freckles
  * cumulative UV exposure
  Measurements will be assessed with questionnaire from about 150 participants.

OTHER OUTCOMES:
Transplantation history | 1 year
  Measurements will be assessed with questionnaire from about 150 participants.

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Hofbauer, Prof MD, Principal Investigator — University Hospital Zurich, Division of Dermatology
Locations (1):
- Universitätsspital Zürich, Zurich, Canton of Zurich, Switzerland